CLINICAL TRIAL: NCT07029594
Title: Interest of Thermal Spa Treatment in Improving ENT-Related Quality of Life in Patients With Primary Ciliary Dyskinesia
Brief Title: Thermal Spa Treatment and Improvement of Primary Ciliary Dyskinesia
Acronym: CANDY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Collaborators: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2022/87
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Primary Ciliary Dyskinesia
MeSH Terms: conditions — Ciliary Motility Disorders | interventions — Balneology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Groupe A (Experimental): Group starting with thermal spa treatment
  Interventions: Other: balneotherapy
- Group B (Experimental): Group starting with prophylactic treatment
  Interventions: Other: balneotherapy

INTERVENTIONS:
Other: balneotherapy — Specific procedures performed during the 3-week spa therapy
  Thermal Treatments (Number of sessions)
  Individual nasal irrigation (18) Sonic aerosol therapy (18) Simple aerosol therapy (18) Individual inhalation therapy (18)
  Administered by a licensed physiotherapist
  Individual respiratory rehabilitation and bronchial drainage (18)
  Administered by a spa physician Tubo-tympanic insufflation (9) Sinus lavage using the Proëtz displacement method 9

SUMMARY:
The goal of this clinical trial is to evaluate whether a 3-week thermal spa treatment can improve quality of life and reduce ENT (ear, nose, and throat) symptoms in adults with Primary Ciliary Dyskinesia (PCD). PCD is a rare, chronic condition that affects the airways and often leads to persistent sinus, ear, and lung infections.

The main questions the study aims to answer are:

Does spa therapy improve ENT-related symptoms and daily quality of life?

Does it help reduce the frequency of infections and the need for antibiotics?

Are there improvements in hearing and lung function?

In this study, participants will be randomly assigned to one of two groups:

Group A will begin with a 3-week spa treatment, followed by regular checkups for 6 months.

Group B will start with standard care for 6 months, then receive the spa treatment and follow-up evaluations for another 6 months.

All participants will:

Undergo ENT and lung function evaluations (questionnaires, hearing tests, nasal swabs, spirometry)

Visit one of two spa centers for a 3-week treatment period (without hospital stay)

Be followed regularly over several months for checkups and tests

Researchers will compare participants' symptoms and test results before and after the spa treatment to determine its benefits.

Potential benefits:

Participants may experience relief from nasal symptoms, fewer respiratory infections, improved hearing and breathing, and an overall better quality of life.

Potential risks:

There is a small risk of infection from a new germ or a mild, short-term flare-up of chronic symptoms (called a "thermal reaction") that can occur during spa therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Primary Ciliary Dyskinesia (PCD) based on electron microscopy analysis of ciliary ultrastructure and/or genetic testing (i.e., two unambiguous mutations in genes known to be involved in PCD, particularly in cases with normal ciliary ultrastructure [~20% of patients], atypical ultrastructural findings, or suggestive symptoms in a family with a known causal gene).
* Age over 18 years.
* Stable maintenance treatment for at least 1 month prior to inclusion.
* Performance Status (PS) ≤ 1.
* Patient has received the study information sheet and signed the informed consent form.
* Patient has valid health insurance coverage.

Exclusion Criteria:

* Participation in a thermal spa treatment within the past year.
* Severe general health deterioration or debilitating conditions.
* Severe or recent heart failure.
* Labile hypertension.
* Venous insufficiency or deep vein thrombosis within the past 3 months.
* Recent unhealed fracture.
* Unhealed skin lesions (wounds, pressure sores, eczema).
* Contagious or progressive diseases.
* Recent cancer (less than 5 years).
* Ongoing or recent (within the past month) pulmonary or ENT exacerbation at inclusion.
* Ongoing treatment with immunomodulatory or immunosuppressive drugs (due to the risk of potentially severe opportunistic infections).
* Ongoing or recent (within the past month) extra-respiratory or ENT infectious flare-up.
* Positive pre-cure bacteriological testing for multidrug-resistant Pseudomonas aeruginosa, MRSA, Mycobacterium abscessus, or other multidrug-resistant pathogenic bacteria.
* Fever > 38.5°C.
* Recently worsened dyspnea (< 1 month).
* History of serious adverse effects or intolerance during a previous thermal spa treatment.
* Participation in another clinical trial with an exclusion period.
* Considered a vulnerable person, as defined by Articles L1121-5 to L1121-8 of the French Public Health Code:

Pregnant women, women in labor, and breastfeeding mothers.

Individuals deprived of liberty by judicial or administrative decision, or those hospitalized without consent under Articles L.3212-1 and L.3213-1 (excluding Article L.1121-8), and persons admitted to a healthcare or social institution for reasons other than research.

Adults under legal protection or unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2026-12-05 (Estimated); Study Completion 2027-05-05 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 6 months
  The primary objective of this study is to evaluate whether a thermal spa treatment leads to a significant improvement in quality of life, as well as in respiratory and auditory symptoms, in patients with primary ciliary dyskinesia. The primary outcome will be the improvement, after spa therapy, of a validated French-language ENT quality of life score specifically designed to assess functional complaints and quality of life in patients with conditions affecting the nasal passages.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire de la Face et du Cou, Nice, France